CLINICAL TRIAL: NCT02240303
Title: Central and Peripheral Mechanisms Predicting Clinical Pain and Physical Performance in Older Adults
Brief Title: Pain, Brain and Mobility Study
Acronym: PBAM
Status: Withdrawn | Type: Observational
Why Stopped: Consolidated study with another protocol
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 201400471
Record Dates: First submitted 2014-09-02; First posted 2014-09-15 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Clinical Pain; Brain and Mobility Changes
Keywords: pain; mobility; brain; cognition
MeSH Terms: conditions — Pain | interventions — Physical Functional Performance; Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Pain Group: Participants that experience chronic pain will have the following procedures performed: A sensory assessment called quantitative sensory testing or QST that will assess in detail your ability to feel sensations due to touch, vibration, and changes in temperature on the skin; Pressure sense will be produced by a device that will be pressed against the skin for several seconds; Pinprick pressure will be applied to determine if the pain can be rated; a Physical Performance test will be performed; and an magnetic resonance imaging (MRI) will be done. In addition, blood sample, blood pressure, heart rate, and skin temperature will be taken during the procedures.
  Interventions: Procedure: Quantitative Sensory Testing (QST); Procedure: Physical Performance; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Blood Sample
- No Chronic Pain Group: Participants that do not experience chronic pain will have the following procedures performed: A sensory assessment called quantitative sensory testing or QST that will assess in detail your ability to feel sensations due to touch, vibration, and changes in temperature on the skin; Pressure sense will be produced by a device that will be pressed against the skin for several seconds; Pinprick pressure will be applied to determine if the pain can be rated; a Physical Performance test will be performed; and an magnetic resonance imaging (MRI) will be done. In addition, blood sample, blood pressure, heart rate, and skin temperature will be taken during the procedures.
  Interventions: Procedure: Quantitative Sensory Testing (QST); Procedure: Physical Performance; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Blood Sample

INTERVENTIONS:
Procedure: Quantitative Sensory Testing (QST) — Participants in both groups will have a sensory assessment called quantitative sensory testing or QST that will assess in detail your ability to feel sensations due to touch, vibration, and changes in temperature on the skin.
Procedure: Physical Performance — Participants in both groups will have a Physical Performance test.
Procedure: Magnetic Resonance Imaging (MRI) — Participants in both groups will have an magnetic resonance imaging (MRI).
Procedure: Blood Sample — Participants in both groups will have blood samples taken.

SUMMARY:
The aim of this project will be to document the central and peripheral mechanisms, which may predict clinical pain characteristics and associated physical performance in older adults. Although chronic pain is common among older adults, there is limited understanding on the processing of pain and the mechanisms by which it affects physical function in these individuals. The first aim of this study will be to examine predictors of clinical pain in older adults. These will include a comprehensive somatosensory assessment battery including mechanical and thermal detection and pain thresholds in older adults with and without chronic pain. The investigators will also assess basal cognitive and physical function to determine their associations with chronic pain. Finally, brain structure and function will be assessed in these older adults with and without pain.

DETAILED DESCRIPTION:
The purpose of this research study is to learn more about how pain in older individuals changes the brain and impacts a person's mobility and function. Pain is influenced by biology (like hormones), psychology (thoughts and feelings), and habits (like sleep or exercise) that may make older adults more likely to have higher or lower levels of pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Willingness to participate in all study procedures
* Cognitively intact as defined by 3MS score > 80

Exclusion Criteria:

* Failure to provide informed consent;
* Contraindications to MRI, such as claustrophobia, heart pacemaker / defibrillator, heart valve prosthesis, aneurysm clip, metallic stent, neurostimulation system, cochlear implants or inner ear prosthesis, insulin pump or other infusion pump, metal slivers in the orbital area/eye socket
* Active treatment for cancer or history of cancer in the past year
* Severe cardiac disease, including New York Heart Association (NYHA) Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest or stroke, use of a cardiac defibrillator, or uncontrolled angina;
* Previous stroke with upper and/or lower extremities involvement within the last 6 months
* History of life-threatening cardiac arrhythmias, stroke, severe Parkinson's disease or severe neurological disorders likely to interfere with physical function
* Renal disease requiring dialysis
* Lung disease requiring steroids
* Inability to reliably rate pain intensity
* Current use of tobacco products
* Uncontrolled hypertension (BP of greater than 150/99 mm Hg)
* Serious systemic disease that restrict normal daily activities
* Neurological problems with significant changes in somatosensory and pain perception at the intended stimulation sites,
* Uncontrolled psychiatric condition (e.g., experiencing symptoms of schizophrenia, bipolar disorder, etc.) or hospitalization within the preceding year for psychiatric illness
* Daily use of narcotic medication
* Lower extremity amputation
* Uncontrolled diabetes (self-reported medication use and/or HA1C value)
* A known diagnosis of dementia
* Inability to communicate because of severe hearing loss or speech disorder;
* Severe visual impairment, which would preclude completion of the assessments and/or intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Brain magnetic resonance imaging (MRI) | Baseline and 12 months later
  Differences in the MRI on the brain scans of participants with greater pain severity

SECONDARY OUTCOMES:
Inflammatory markers in blood samples | Baseline
  To test the markers of pro-inflammatory (IL-1b, tumor necrosis factor (TNF-a)) and anti-inflammatory (IL-4, IL-10) with participants more sensitive to pain than the ones less sensitive to pain.

OTHER OUTCOMES:
Mobility (gait speed) | Baseline and 12 months
  Inverse dynamics will be used to calculate gait speed.

CONTACTS AND LOCATIONS:
Overall Officials: Yenisel Cruz-Almeida, MSPH, PhD, Principal Investigator — University of Florida